CLINICAL TRIAL: NCT04584996
Title: CIRcular and Non-coding RNAs as Clinically USeful Biomarkers in Pancreaticobiliary Cancers
Acronym: CIRCUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 277406
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Pancreatic Cancer; Biliary Tract Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pancreatic cancer: Patients being evaluated at MDT for suspected Pancreatic Ductal Adenocarcinoma (PDAC), via radiological test (e.g. endoscopic ultrasound (EUS), endoscopic retrograde cholangiography (ERCP), cross-sectional imaging), serum tumour marker (i.e. CA 19-9), or other diagnostic procedure
- Control: Patients diagnosed and/or due to undergo surgery for benign pathology (e.g. gallstones, chronic pancreatitis, etc); or patients with a diagnosis of a pre-malignant lesion (e.g. pancreatic intraductal papillary mucinous neoplasm); Pancreatic Neuroendocrine Tumour, or a Biliary Tract Cancer (i.e. cholangiocarcinoma; gallbladder cancer; ampullary cancer)

SUMMARY:
1. Define the circRNA expression profile in PDAC and identify dysregulated circRNA candidates. These will be validated in further tissue samples.
2. Evaluate candidate circRNA Expression in blood (plasma samples) as a clinically relevant diagnostic biomarker; expanding on the primary objective to include other diagnostic features such as specificity, area under the receiver operator curve, positive predictive value and negative predictive value.
3. Explore the expression of candidate circRNAs and related molecules in patient biomaterials (including tissue, blood, bile and biopsy samples) as biomarkers for diagnosis; prognostication; association with clinico-pathologic features and survival outcomes; and their ability to predict/monitor treatment response e.g. surgery and/or chemotherapy.
4. Utilise computer-based analyses to describe the theoretical interactions of candidate circRNAs within the full complement of RNA and related molecules produced by the tumour cells, called the 'transcriptome', in human PDAC.

DETAILED DESCRIPTION:
This first step of this project is a 'discovery experiment' to describe the expression profiles of 8 PDAC tissue samples compared to controls; with subsequent validation of candidate circRNAs:

8 paired samples of PDAC tumour tissue and associated normal pancreatic tissue will be collected at the time of surgery (after the pancreatic tumour is resected). The expression levels of circRNAs will be profiled and the most significantly dysregulated candidate circRNAs will be chosen (also considering other datasets and the current literature in this decision).

The second step of this project is a prospective non-interventional observational cohort study to investigate these candidate circRNAs further:

The expression of these candidate circRNAs expression levels will be measured longitudinally throughout the clinical timeline of patients with PDAC in blood samples; and in bile, tissue and biopsy samples (when this is safely available after clinical sampling and without additional investigations). This will be compared against control patients with benign biliary disease and other biliary tract cancers. These controls would only be available for blood tests and, if undergoing cholecystectomy, bile. Blood tests will be taken alongside clinical bloods or after anaesthesia for surgical procedures, bile will be taken after removal of the gallbladder for gallstone disease when this is in excess to clinical requirements.

The ability of each circRNAs as a diagnostic, prognostic and predictive biomarkers will be described and compared to CA 19-9 (the only biomarker that is currently widely accepted in PDAC). This will first be considered in blood samples and then other patient biomaterials.

The final part of the project will be to undertake both computer and laboratory evaluation of candidate circRNAs in order to propose a its molecular relationships and how this may explain and associations described.

A Bioinformatical review will give the ability to computationally determine the miRNA-binding capabilities of candidate circRNAs, and the downstream mRNAs regulated. Gene-ontology and KEGG pathway enrichment-analyses of the differentially expressed genes will allow a global-view of the transcriptome under circRNA regulation in PDAC.

ELIGIBILITY:
Inclusion Criteria:

* Participants capable of giving informed consent
* Aged >18 years

Exclusion Criteria:

* Unwilling or unable to provide written informed consent
* Non-English speaking
* Known to be pregnant
* Aged <18 years
* Known diagnosis of HIV or Hepatitis B/C virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being evaluated at MDT for suspected Pancreatic Ductal Adenocarcinoma (PDAC), via radiological test (e.g. endoscopic ultrasound (EUS), endoscopic retrograde cholangiography (ERCP), cross-sectional imaging), serum tumour marker (i.e. CA 19-9), or other diagnostic procedure
Sampling Method: Non-Probability Sample
Enrollment: 186 (Estimated)
Dates: Start 2020-10-04 (Actual); Primary Completion 2021-10-05 (Estimated); Study Completion 2023-11-05 (Estimated)

PRIMARY OUTCOMES:
circRNAs for diagnosis | 12 months
  To identify a plasma circRNA 'signature' able to diagnose Pancreatic Ductal Adenocarcinoma (PDAC) with superior sensitivity than serum CA 19-9

SECONDARY OUTCOMES:
Describe circRNAs expression profile | 12 months
  Define and validate the circRNA expression profile in PDAC and identify dysregulated circRNA candidate(s).
Diagnostic features of blood circRNAs | 12 months
  Evaluate candidate circRNA expression in blood (plasma) as a clinically relevant diagnostic biomarker; expanding on the primary objective to include other diagnostic features, such as specificity, area under the receiver operator curve, positive predictive value and negative predictive value
circRNAs in other biomaterials | 30 months
  Explore the expression of candidate circRNAs, and related molecules, in patient biomaterials (including tissue, blood, bile and biopsy samples) as biomarkers for diagnosis; prognostication; association with clinico-pathologic features and survival outcomes; and their ability to predict/monitor treatment response (i.e. surgery and/or chemotherapy).
Bioinformatics | 18 months
  tilise computer-based analyses to describe the theoretical interactions of candidate circRNAs within transcriptome in human PDAC.

CONTACTS AND LOCATIONS:
Overall Officials: C A Limb, MBBS MRes, Principal Investigator — The Royal Surrey NHS Foundation Trust
Locations (1):
- Royal Surrey County Hospital, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No